CLINICAL TRIAL: NCT03692039
Title: Comparison of Postoperative Pain After Root Canal Instrumentation Using M-Pro and ProTaper Next in Molars With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Comparison Between M-Pro and ProTaper Next
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Essam Othman Ibrahim, Resident at Endodontic department Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-33
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Intervention Model Description: Blocks of 4 are generated on a Microsoft Excel sheet where the intervention and control are denoted A & B and randomly distributed. The table is kept with the assistant supervisor.
Who Masked: Participant
Masking Description: After the operator find an eligible participant, a phone call is made to the assistant supervisor to confirm the patient eligibility then to assign the participant to either group according to the generated random sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-pro files (Experimental): Instrumentation using M-pro files in rotating motion
  Interventions: Procedure: M-pro files in rotating motion
- ProTaper Next files (Active Comparator): Instrumentation using ProTaper Next files in rotating motion
  Interventions: Procedure: ProTaper Next files in rotating motion

INTERVENTIONS:
Procedure: M-pro files in rotating motion — An endodontic file that has controlled memory properties
  Arms: M-pro files
Procedure: ProTaper Next files in rotating motion — An endodontic file that has an off center mass of rotation
  Arms: ProTaper Next files

SUMMARY:
Comparing the postoperative pain resulting after mechanical instrumentation using M-pro files versus that resulting after using ProTaper Next rotary files in lower molar with symptomatic Irreversible pulpitis molars.

DETAILED DESCRIPTION:
Lower molars with symptomatic Irreversible pulpitis molars are selected according to the eligibility and exclusion criteria and patients are then randomized to receive treatment either using M-pro Files or ProTaper Next files. Postoperative pain is then assessed using the Numerical Rating scale 6, 12, 24, 48 and 72 hours post-operatively . After completing the treatment, patients will instructed to take placebo if they feel pain and will be asked to provide the quantity of placebo intake until 72 hrs. In case of pain not relieved by placebo, after recording the amount of pain, the patient will be instructed to take an alternative line of pain control (Ibuprofen 400mg tablets every 6 hours). The amount and frequency of Ibuprofen intake will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1- Males or Females.
* 2- Mandibular molar teeth with:

  * Pre-operative sharp pain.
  * Vital response of pulp tissue to cold pulp tester (ethyl chloride spray).
  * Normal periapical radiographic appearance or slight widening in lamina dura using periapical index (PAI) score 1 as normal periapical structures or 2 as small changes in bone structures.

Exclusion Criteria:

* Patients having significant systemic disorders.
* Patients who are allergic to non-steroidal anti-inflammatory drugs.
* Patients with two or more adjacent teeth requiring root canal therapy.
* Teeth that have:

  * Necrotic pulp tissues.
  * Association with swelling or fistulous tract.
  * Acute or chronic peri-apical abscess.
  * Greater than grade I mobility.
  * Pocket depth greater than 5mm.
  * No possible restorability.
  * Previous endodontic treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain assessed with numerical rating scale | Up to 72 hours post-operatively
  0 (none) to 10 (severe) Numerical Pain Rating Scale up to 72 hours post-operatively

SECONDARY OUTCOMES:
Incidence of placebo intake assessed by questioning | Up to 72 hours post-operatively
  Amount of placebo intake up to 72 hours post-operatively
Amount of analgesic intake assessed by counting | Up to 72 hours post-operatively
  Number of analgesic tablets up to 72 hours post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kocak MM, Cicek E, Kocak S, Saglam BC, Furuncuoglu F. Comparison of ProTaper Next and HyFlex instruments on apical debris extrusion in curved canals. Int Endod J. 2016 Oct;49(10):996-1000. doi: 10.1111/iej.12552. Epub 2015 Oct 12. PMID 26383696
- [Background] Ruddle CJ, Machtou P, West JD. The shaping movement: fifth-generation technology. Dent Today. 2013 Apr;32(4):94, 96-9. No abstract available. PMID 23659098